CLINICAL TRIAL: NCT04955704
Title: Performance Study for InferRead CT Pneumonia.AI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Infervision (Industry)
Collaborators: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Other Study IDs: PNEUMONIA06142021
Record Dates: First submitted 2021-06-22; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: InferRead CT Pneumonia.AI — InferRead CT Pneumonia.AI reads chest CT DICOM images from medical imaging storage devices and triages cases by detecting pneumonia lesions and then flagging suspected cases in the study list. InferRead CT Pneumonia.AI is a tool to assist clinicians and it does not replace the interpretation and diagnosis by clinicians.

SUMMARY:
A retrospective, blineded, multicenter study of the InferRead CT Pneumonia.AI to evaluate the performance in identifying non-contrast chest CT scans containing pneumonia findings.

DETAILED DESCRIPTION:
This is a retrospective, blinded, multicenter study for the InferRead CT Pneumonia.AI. The primary endpoint will evaluate the software's performance in identifying non-contrast chest CT scans containing pneumonia. It will evaluate InferRead CT Pneumonia.AI in terms of sensitivity and specificity with respect to a ground truth, as established by trained thoracic radiologists, in the detection of penumonia. In addition, the study will compare time to notification for the InferRead CT Pneumonia.AI software with respect to the time to notification for the standard of care as established from available radiological reports.

1. To evaluate the performance of InferRead CT Pneumonia.AI.
2. To evaluate the effect of different factors such as CT manufacturer, CT scanning protocols and patient characteristics on the performance of InferRead CT Pneumonia.AI

ELIGIBILITY:
Inclusion Criteria:

1. Non-contrast chest CT DICOM scans
2. Contains both lung lobes
3. Slice thickness is less than 3 mm.

Exclusion Criteria:

1. Incomplete scan or corrupted scan
2. Irregular scanning, increased intrapulmonary density due to insufficient inspiration, and respiratory artifacts affecting the physician's judgment.
3. Altered or absent lung morphology in the postoperative patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This retrospective study will be used to assess the performance of the subject device. The principal investigator will collect DICOM data and relevant clinical information based on the selection criteria. DICOM will be de-identified of PHI and stored in a secure location.
  The validation dataset will contain non-contrast chest CT scans from patients in the United States that are either negative or have confirmed pneumonia (viral or bacterial). Data will come from at least 3 hospitals and cover a variety of data attributes.
Sampling Method: Probability Sample
Enrollment: 423 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | 1/1/2022 - 2/28/2022
  1. The Sensitivity (SE) of InferRead CT Pneumonia.AI is higher than 0.80. H0: YSE ≤ 0.80 HA: YSE > 0.80
  2. The Specificity (SP) of InferRead CT Pneumonia.AI is higher than 0.80. H0: YSP ≤ 0.80 HA: YSP > 0.80

SECONDARY OUTCOMES:
Secondary Endpoint | 1/1/2022 - 2/28/2022
  The Average Per Case Processing Time of InferRead CT Pneumonia.AI is lower than Time-to-open-exam in the standard of care
  H0: Per Case Processing Time ≥ Time-to-open-exam HA: Per Case Processing Time < Time-to-open-exam
  The Average Per Case Processing Time of InferRead CT Pneumonia.AI includes the time to receive the DICOM exam and the shows AI results on the studylist. The standard of care time-to-open-exam is defined as the time from the initial scan of the patient to the time when the radiologist first opens the exam for review.